CLINICAL TRIAL: NCT06808633
Title: Efficacy of Direct Selective Laser Trabeculoplasty in Clinical Practice in Patients with Glaucoma
Status: Recruiting | Type: Observational
Sponsor: Clínica Rementería (Other)
Responsible Party: Sponsor
Other Study IDs: 25/033-E
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma
Keywords: glaucoma; direct selective laser trabeculoplasty
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study participants: Age over 18 years Diagnosis of open angle glaucoma instudy eye and scheduled for both eyes being treated after bilateral laser indication. The diagnosis of glaucoma will be based on the presence of optic nerve damage that is compatible with glaucoma in the absence of any other cause that could have produced this damage, with an IOP value>21 mmHg.

SUMMARY:
Prospective, single-arm, single-center, non-randomized, non-comparative study including naïve patients attending our center diagnosed with glaucoma, who have been recommended treatment with direct selective laser trabeculoplasty (DSLT) by their ophthalmologist and who are under no hypotensive medication. DSLT treatment will be performed with the Voyager DSLT system; it will consist of the application of 120 laser pulses of preset 3 ns and a preset 400 μm spot size, with an energy of 1.8 mJ delivered to the limbus through a full 360 degrees.

The study will evaluate the effect of DSLT on intraocular pressure (IOP). Baseline IOP will be the IOP measured with Goldman applanation tonometry by the investigator on the day of treatment, prior to the application of DSLT. Patients will be seen one week (±2 days), one month (±7 days), three months (±15 days), six months (±30 days) and 12 months (±40 days) after DSLT treatment. In each of these visits, the attending ophthalmologist will measure IOP with Goldmann applanation tonometry and record the presence of any relevant ocular signs and query patients regarding potential adverse events. The study´s main end-point will be percentage reduction in IOP six months after DSLT compared to baseline.

ELIGIBILITY:
Inclusion Criteria: • Age over 18 years

• Diagnosis of open angle glaucoma in eye study and scheduled for both eyes being treated after bilateral laser indication. The diagnosis of glaucoma will be based on the presence of optic nerve damage that is compatible with glaucoma in the absence of any other cause that could have produced this damage, with an IOP value>21 mmHg.

Exclusion Criteria:

* Patients diagnosed with uveitis, angle closure or congenital glaucoma.
* Presence of anterior peripheral synechiae
* Patients unable to complete three, six- and 12-months follow-up.
* Patients having undergone intraocular surgery, save for uneventful phacoemulsification (performed at least 6 months prior to inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with open angle glaucoma in study eye and scheduled for both eyes being treated after bilateral laser indication.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Percentage change in IOP six months after DSLT compared to baseline. | 6 months after DLST application
  Percentage change in IOP six months after DSLT compared to baseline.

SECONDARY OUTCOMES:
Percentage change in washed-out IOP 3 and 12 months after DSLT compared to baseline. | 12 months
  Percentage change in washed-out IOP 3 and 12 months after DSLT compared to baseline.
Mean washed-out IOP change 3, 6 and 12 months after DSLT compared to baseline. | 12 months
  Mean washed-out IOP change 3, 6 and 12 months after DSLT compared to baseline.
Proportion of participants with at least 20% reduction in washed-out IOP from baseline at 3, 6 and 12 months. | 12 months
  Proportion of participants with at least 20% reduction in washed-out IOP from baseline at 3, 6 and 12 months.
Percentage of patients using hypotensive topical treatment after DSLT at 3, 6, and 12 months | 12 months
  Percentage of patients using hypotensive topical treatment after DSLT at 3, 6, and 12 months
Mean number of medications 3, 6 and 12 months after DSLT (accounting for those on no medications as well when calculating the average). | 12 months
  Mean number of medications 3, 6 and 12 months after DSLT (accounting for those on no medications as well when calculating the average).

OTHER OUTCOMES:
Glaucoma Quality of Life-15 Questionnaire at 12 months after DSLT. | 12 months
  Glaucoma Quality of Life-15 Questionnaire at 12 months after DSLT. It consists of 15 questions asking about patients difficulty for performing everyday tasks, which the patient must grade from 1 to 5, with 1 being that patient has no difficulty performing the task and 5 that he has severe diificulties. Values range from 15 (no difficulties for any activity) to 45 (has severe difficulties for performing all activities)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Rementería, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Age, gender, baseline IOP, severity of glaucoma, IOP at each follow-up visit, need for glaucoma medications
Supporting Information: CSR
Time Frame: At the end of study (expected winter 2026) and for five years
Access Criteria: Data deposited in a dataset repository, accessed by identified researchers